CLINICAL TRIAL: NCT00001618
Title: Bronchoscopy in Patients With Pulmonary Diseases and Research Volunteers
Brief Title: Segmental Bronchoalveolar Lavage
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970022; 97-H-0022
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08-31

CONDITIONS: Asthma; Pulmonary Fibrosis
Keywords: Cystic Fibrosis; Healthy Volunteers; Asthma; Normal Volunteer; Chronic Lung Disease
MeSH Terms: conditions — Asthma; Pulmonary Fibrosis; Cystic Fibrosis

SUMMARY:
Bronchoalveolar lavage (BAL) is a diagnostic and therapeutic procedure conducted by placing a small fiberoptic scope into the lung of a patient, and injecting sterile water (saline) into the lung and removing the fluid. The sterile solution removed contains secretions, cells, and protein from the lower respiratory tract. This sample can be analyzed to provide more information about possible disease processes going on in the lungs.

This protocol will be used to perform BAL, bronchial brushing, and bronchial wall biopsy in normal volunteers and patients with pulmonary disease. The samples collected during the study will be used to examine biochemical processes in the lung that may contribute to lung disease

DETAILED DESCRIPTION:
This protocol proposes to perform bronchoalveolar lavage, bronchial brushing and bronchial wall biopsy in research volunteers and in patients with pulmonary disease to evaluate the cellular components of normal and diseased lungs. This research study will help to improve our understanding of pathogenic mechanisms in the lung during progression of pulmonary disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients and research volunteers will be accepted for bronchoscopy and bronchoalveolar lavage only if their heath status will not be compromised by the procedure. Examples of disease that may be studied under this protocol include alpha-1 antitrypsin deficiency; lymphangioleiomyomatosis and the cystic lung disease; pulmonary fibrosis; and sarcoidosis.

EXCLUSION CRITERIA:

Patients or research volunteers with abnormalities that contraindicate, or increase the risk of, fiberoptic bronchoscopy and bronchoalveolar lavage, including a history of allergy to atropine, lidocaine, or other topical anesthetics or premedications; FEV(1) less than 0.8 liters; PaO(2), on supplemental 02, of less than 70 mmHg or PaCO(2) greater than 45 mmHg; presence of uncorrected clotting disorder, uncontrolled hypertension, significant cardiac disease, renal or liver failure; metastatic disease; hematologic disorders such as severe anemia (hemoglobin less than or equal to 7 g/ml), granulocytopenia, or platelet disorders.

Patients or research volunteers with a positive serum test for human immunodeficiency virus or hepatitis B or C. The rationale for excluding participation on the basis of HIV seropositivity is because of the known effects of HIV on the lungs.

Patients or research volunteers who are pregnant or lactating.

Patients or research volunteers incapable of giving informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 1996-11-18; Study Completion 2018-08-31

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Elston WJ, Whittaker AJ, Khan LN, Flood-Page P, Ramsay C, Jeffery PK, Barnes NC. Safety of research bronchoscopy, biopsy and bronchoalveolar lavage in asthma. Eur Respir J. 2004 Sep;24(3):375-7. doi: 10.1183/09031936.04.00063003. PMID 15358694
- [Background] Chapman JT, Mehta AC. Bronchoscopy in sarcoidosis: diagnostic and therapeutic interventions. Curr Opin Pulm Med. 2003 Sep;9(5):402-7. doi: 10.1097/00063198-200309000-00011. PMID 12904711
- [Background] Jarjour NN, Peters SP, Djukanovic R, Calhoun WJ. Investigative use of bronchoscopy in asthma. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):692-7. doi: 10.1164/ajrccm.157.3.9705020. PMID 9517577